CLINICAL TRIAL: NCT04699539
Title: Recurrence-pattern-based Volume Versus Conventional-volume Stereotactic Body Radiation Therapy in Locally Advanced Pancreatic Cancer: an Open-label, Randomized, Phase 2 Trial
Brief Title: Different Patterns of Target Delineation in SBRT for Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Director, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Changhai Hospita
Record Dates: First submitted 2020-11-09; First posted 2021-01-07 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Treatment
Keywords: SBRT; Locally Advanced Pancreatic Cancer; Target Delineation
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): A conventional-volume stereotactic body radiation therapy following gemcitabine and nab-paclitaxel
  Interventions: Radiation: SBRT; Drug: Chemotherapy
- Arm B (Experimental): A recurrence-pattern-based-volume stereotactic body radiation therapy following gemcitabine and nab-paclitaxel
  Interventions: Radiation: SBRT; Drug: Chemotherapy

INTERVENTIONS:
Radiation: SBRT — A conventional-volume stereotactic body radiation therapy: planning target volume should include gross tumor volume with a uniform 3mm margin in all directions.
  A recurrence-pattern-based volume stereotactic body radiation therapy: planning target volume should include gross tumor volume with a 3mm margin in the anterior and lateral directions, 10mm margin in the cranial and caudal directions that should cover the full circumstance of celiac artery and superior mesenteric artery, 15mm in the posterior direction that should cover the retroperitoneal space.
  The prescribed dose of PTV varies from 30-50Gy/5-6f.
Drug: Chemotherapy — Gemcitabine (1000mg/m2，d1, 8) + albumin-bound paclitaxel (125mg/m2，d1, 8) , repeat every 3 weeks for 6 cycles

SUMMARY:
The purpose of this study is to compare the efficacy and safety of a recurrence-pattern-based-volume versus conventional-volume stereotactic body radiation therapy for locally advanced pancreatic cancer, so as to determine whether the target delineation method based on recurrence pattern can obtain better survival benefits.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically verified pancreatic adenocarcinoma
* Imaging examinations confirmed locally advanced pancreatic cancer
* No previous radiotherapy, chemotherapy, immunotherapy or targeted therapy
* ECOG of 0 to1
* Age of 18 years or older
* Adequate bone marrow function, defined as: Absolute neutrophil count (ANC) ≥ 1.5×10^9 cells/L, leukocyte count≥ 3.5×10^9 cells/L, platelets ≥ 70×10^9 cells/L, hemoglobin ≥ 8.0 g/dl
* Adequate liver and renal, defined as: Albumin > 2.5 g/dL, total bilirubin < 3 mg/dL, creatinine < 2.0 mg/dL, AST<2.5 × ULN (Upper Limit of Normal) (0-64U/L), ALT<2.5 × ULN (0-64U/L)
* Adequate blood clotting function, defined as: international normalized ratio (INR) < 2 (0.9-1.1)
* Ability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Previously receiving radiotherapy, chemotherapy, immunotherapy or targeted therapy
* Evidences of metastatic disease confirmed by chest CT or PET-CT
* ECOG ≥2
* Age <18 years
* Secondary malignancy
* Abnormal results of blood routine examinations and liver and kidney and coagulation tests
* Patients with active inflammatory bowel diseases or peptic ulcer
* Gastrointestinal bleeding or perforation within 6 months
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
* Medical history of symptomatic congestive heart failure: New York Heart Association Class III to IV
* Medical history of respiratory insufficiency
* Women who are pregnant or breastfeeding
* Participation in another clinical treatment trial
* Inability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-08-16 (Actual); Study Completion 2025-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: A conventional-volume SBRT following gemcitabine and nab-paclitaxel
- Arm B: A recurrence-pattern-based-volume SBRT following gemcitabine and nab-paclitaxel
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 47 | 49
Completed | 47 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 47 | 49 | 96
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [57 to 73] | 63 [58 to 74] | 63.5 [58 to 73.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 26 | 29 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Age, Continuous [Median (Inter-Quartile Range); unit: yerars] | 66 [57 to 73] | 63 [58 to 74] | 63.5 [58 to 73.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 26 | 29 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Participants [Count of Participants; unit: Participants] | 47 | 49 | 96

OUTCOME MEASURES:

1. Primary Outcome: 1-year Progression Free Survival Rate
Description: The proportion of patients without disease progression at one year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 47 | 49
Participants | 9 | 18

2. Secondary Outcome: Treatment-related Adverse Events
Description: Treatment-related adverse events
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 47 | 49
Participants | 45 | 46

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival
Time Frame: 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 47 | 49
months | 7.3 [4.5 to 10.1] | 9.6 [7.3 to 11.9]

4. Secondary Outcome: Overall Survival
Description: Overall Survival
Time Frame: 4 years
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 47 | 49
months | 10.8 [9.7 to 11.9] | 15.2 [11.6 to 18.8]

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 47/47 | 49/49
Serious Adverse Events (participants affected / at risk) | 20/47 | 21/49
Other Adverse Events (participants affected / at risk) | 43/47 | 42/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=47) | Arm B (N=49)
Leukopenia (Blood and lymphatic system disorders) | 10 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 10
Anemia (Blood and lymphatic system disorders) | 3 | 0
Nausea or vomiting (Gastrointestinal disorders) | 6 | 9
Diarrhea (Gastrointestinal disorders) | 2 | 1
Decreased appetite (Gastrointestinal disorders) | 7 | 11
Elevated aspartate aminotransferase (Hepatobiliary disorders) | 8 | 7
Elevated alanine aminotransferase (Hepatobiliary disorders) | 5 | 6
Hypoalbuminemia (Hepatobiliary disorders) | 1 | 0
Weight decreased (Metabolism and nutrition disorders) | 6 | 7
Fatigue (General disorders) | 4 | 9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=47) | Arm B (N=49)
Leukopenia (Blood and lymphatic system disorders) | 36 | 39
Thrombocytopenia (Blood and lymphatic system disorders) | 27 | 30
Anemia (Blood and lymphatic system disorders) | 8 | 5
Nausea or vomiting (Gastrointestinal disorders) | 38 | 36
Diarrhea (Gastrointestinal disorders) | 11 | 14
Decreased appetite (Gastrointestinal disorders) | 39 | 40
Constipation (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Elevated aspartate aminotransferase (Hepatobiliary disorders) | 23 | 26
Elevated alanine aminotransferase (Hepatobiliary disorders) | 22 | 27
Blood bilirubin increased (Hepatobiliary disorders) | 4 | 2
Hypoalbuminemia (Hepatobiliary disorders) | 9 | 5
Weight decreased (Metabolism and nutrition disorders) | 24 | 22
Fatigue (General disorders) | 33 | 37
Fever (General disorders) | 7 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 35 | 33
Peripheral neurotoxicity (Nervous system disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT04699539/Prot_SAP_000.pdf